CLINICAL TRIAL: NCT05110417
Title: Pilot Study of the Efficacy of Pyridostigmine for Reversal of Post Injection Dysphonia Following Botulinum Neurotoxin Laryngeal Chemo-Denervation in Spasmodic Dysphonia
Brief Title: Reversal of Botulinum Neurotoxin Injection Related Dysphonia With Pyridostigmine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Benjamin J Rubinstein, Assistant Professor, Eastern Virginia Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V4.0 28July2021
Record Dates: First submitted 2021-09-14; First posted 2021-11-08 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Dysphonia, Spastic; Dysphonia; Laryngeal Dystonia
Keywords: pyridostigmine; dysphonia; spasmodic dysphonia; Mestinon; botulinum neurotoxin
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Intervention Model Description: This is a pilot study so all 10 participants will be assigned to the pyridostigmine (Mestinon) treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pyridostigmine (Mestinon) (Experimental): Pyridostigmine (Mestinon) will be assigned to patients in this arm.
  Interventions: Drug: Pyridostigmine Bromide 60 Milligrams (mg)

INTERVENTIONS:
Drug: Pyridostigmine Bromide 60 Milligrams (mg) — One tablet will be provided to patients during the second visit.
  Other Names: Amneal Pharmaceuticals Pvt. Ltd.; Serial Number: 1000462308

SUMMARY:
The purpose of this study is to evaluate the effects of pyridostigmine (Mestinon) on patient vocal outcomes after undergoing laryngeal botulinum neurotoxin (BoNT) injections, which is a standard treatment for spasmodic dysphonia. Pyridostigmine (Mestinon) has been used for treatment of BoNT overdose, and it is our hope that it will be beneficial in the management of post BoNT breathy phase.

DETAILED DESCRIPTION:
The study will enroll 10 subjects and will involve 1 clinic visit with two sessions over 2 hours.

Participants' voices will then be analyzed via sentence/passage reading, sustained vowel holding, maximum phonation time, as well as subjective ratings of effort. During the second clinic visit, participants will then be administered one 60mg tablet of pyridostigmine (Mestinon) orally, and asked to return to the clinic in 2 hours, when Mestinon has reached peak plasma concentration. Upon returning, participants will repeat the vocal analysis and results will be evaluated for any change in outcome.

Patients who are pregnant, lactating, or have kidney or heart disease should not participate.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females Aged 21-100
* Scheduled for Botulinum Neurotoxin (BoNT) Treatment for Spasmodic Dysphonia (SD)

Exclusion Criteria:

* Subjects who are Pregnant or Lactating
* Subjects with Compromised Renal or Cardiac Function
* Subjects with Spasmodic Dysphonia with Superimposed Vocal Tremor

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Rainbow Passage Reading Pre- and Post-Pyridostigmine (Mestinon) | 15 Minutes
  This pilot study aims to evaluate the efficacy of pyridostigmine (Mestinon) to improve vocal outcomes following laryngeal chemo-denervation with botulinum neurotoxin injection which is a standard of care treatment of adductor spasmodic dysphonia. One of the outcome measures used will be the Rainbow Passage reading. A comparison between pre-pyridostigmine reading and post-pyridostigmine reading will be performed to meet this outcome measure.
CAPE-V Pre- and Post-Pyridostigmine (Mestinon) | 15 Minutes
  This pilot study aims to evaluate the efficacy of pyridostigmine (Mestinon) to improve vocal outcomes following laryngeal chemo-denervation with botulinum neurotoxin injection which is a standard of care treatment of adductor spasmodic dysphonia. Another outcome measurement used will be the Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V). A comparison between the pre-pyridostigmine evaluation of the CAPE-V and post-pyridostigmine evaluation of the CAPE-V will be performed to meet this outcome measure.
Glottal Function Index Pre- and Post-Pyridostigmine (Mestinon) | 15 Minutes
  This pilot study aims to evaluate the efficacy of pyridostigmine (Mestinon) to improve vocal outcomes following laryngeal chemo-denervation with botulinum neurotoxin injection which is a standard of care treatment of adductor spasmodic dysphonia. Another primary outcome measure being assessed is the glottal function index (GFI). A comparison between the pre-pyridostigmine GFI and post-pyridostigmine GFI will be performed to meet this outcome measure. Score is ranked from 0 to 5. The lower the GFI score indicates fewer problems/effort.
Adapted Borg Scale Pre- and Post-Pyridostigmine (Mestinon) | 15 Minutes
  This pilot study aims to evaluate the efficacy of pyridostigmine (Mestinon) to improve vocal outcomes following laryngeal chemo-denervation with botulinum neurotoxin injection which is a standard of care treatment of adductor spasmodic dysphonia. Another primary outcome measure being assessed is the adapted Borg scale. A comparison between the pre-pyridostigmine scale rating and the post-pyridostigmine scale rating will be performed to meet this outcome measure. The scale is ranked from 0 to 10. The higher the number indicates more effort in the tasks while a lower number indicates less effort.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Rubinstein, MD, Principal Investigator — Eastern Virginia Medical School Department of Otolaryngology - Head and Neck Surgery
Locations (1):
- Eastern Virginia Medical School Ear, Nose, and Throat Surgeons, Norfolk, Virginia, United States